CLINICAL TRIAL: NCT05029401
Title: Ibogaine to Determine Maximum Tolerated Dose (MTD) or Treat-to-Target Dose (TTD) for the Evaluation of Efficacy and Safety
Brief Title: A Study of Oral Ibogaine in Opioid Withdrawal
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: atai Therapeutics, Inc. (Industry)
Collaborators: MAC Clinical Research (Other); ERT: Clinical Trial Technology Solutions (Other); Hammersmith Medicines Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMX-IB-201
Record Dates: First submitted 2021-05-13; First posted 2021-08-31 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Opiate Withdrawal Syndrome
Keywords: Opioid withdrawal symptoms; abrupt opioid discontinuation; opioid detoxification; opioid use disorder; substance use disorder
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: The initial Stage 1 (phase 1) design was an open label study. Following review of data from the first cohort in Stage 1, an additional 6 subjects will be recruited into Cohort 1 and the protocol has been amended to implement a multi-centre, single-blind placebo-controlled assessment of QTcF and individualized heart rate correction modeling of QTcI.
  Following baseline evaluations each subject receives placebo (Day 1) followed by ibogaine (Day 2), serving as his or her own control. In addition, data is collected from the baseline assessments (Day -1) to assess QT/RR diurnal variability under normal conditions and in response to autonomic stimulus (i.e. postural changes).
  Stage 2 (phase 2a) is a double-blind, placebo-controlled, parallel group design targeting opioid-dependent patients to receive a single dose of the DMX-1002 or placebo for medically supervised opioid withdrawal.
Who Masked: Participant, Investigator
Masking Description: Stage 1 (phase 1) of the study is single-blind (participant blinded); patients receive one initial dose of placebo, followed by one dose of IMP on the next day, and thereby serve as their own controls.
  Stage 2 (phase 2a) is double-blinded. Patients will be randomized to receive either the IMP or placebo as a single dose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single dose IMP (DMX-1002) (Experimental): Stage 1 (single blind, placebo controlled): initial dose of placebo, followed by treatment at one of 4 ascending dose levels of IMP (3, 6, 9 or 12 mg/kg)
  Stage 2 (blinded): MTD/TTD established in Stage 1 vs placebo (proof of concept)
  Interventions: Drug: DMX-1002; Drug: Placebo
- Matching Placebo (Placebo Comparator): Placebo using capsules identical to the IMP (DMX-1002)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DMX-1002 — Investigation of the safety, tolerability and pharmacokinetics (PK) in healthy volunteers (Stage 1 - single blind), and the efficacy, safety, tolerability and PK in opioid-dependent patients (Stage 2 - double blind)
  Other Names: Ibogaine Hydrochloride
  Arms: Single dose IMP (DMX-1002)
Drug: Placebo — Matching placebo to the IMP (DMX-1002)
  Other Names: Microcrystalline cellulose

SUMMARY:
Study DMX-IB 201 is a Phase 1/2a study of ibogaine consisting of an initial single ascending dose escalation stage to determine the maximum tolerated dose (MTD) or treat-to-target dose (TTD) in healthy volunteers, followed by a randomized, double-blind, placebo-controlled proof of concept stage to demonstrate the efficacy, safety and tolerability of the selected dose in opioid-dependent patients who seek medically supervised opioid withdrawal

DETAILED DESCRIPTION:
Detailed description restricted as elements of this trial are part of a Phase 1 clinical trial.

ELIGIBILITY:
Important Inclusion Criteria for both Stages 1 and 2:

* Males and females between 18 years and 55 years of age.
* For Stage 1, healthy volunteers; recreational opioid use is allowed but not required for inclusion in the study.
* For Stage 2, opioid-dependent subjects (DSM-IV) seeking medically supervised opioid withdrawal and presenting with an OOWS score ≥ 5 on Day 1, prior to dosing.
* Self-report of at least 1 prior positive hallucinogen drug experience that included a meaningful altered state of consciousness. Hallucinogenic substances can include psilocybin, LSD, MDMA or other classic hallucinogens.
* Females that are not of child-bearing potential as defined within the protocol.
* Males who agree to use 1 of the acceptable contraceptive regiments and not to donate sperm from the first study drug administration to at least 90 days after the last drug administration or who are unable to procreate (as defined within the protocol).
* For Stage 1, negative urine tests for drugs of abuse (opiates, benzodiazepines, amphetamines, cannabinoids, cocaine, barbiturates, and phencyclidine), and CNS (central nervous system) prescription drugs (SSRIs [selective serotonin reuptake inhibitors], SNRIs [serotonin-norepinephrine reuptake inhibitors], mood stabilizers) both at screening and within approximately 7 days prior to dosing, and negative alcohol test.
* For Stage 2, negative blood and urine tests for methadone, buprenorphine, mitragynine, non-opioid drugs of abuse (benzodiazepines, amphetamines, cannabinoids, cocaine, barbiturates, and phencyclidine), and CNS prescription drugs (SSRIs, SNRIs, mood stabilizers) both at screening and within approximately 7 days prior to dosing, and negative breath alcohol test at Day -1.
* Negative serology test result for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen, hepatitis C virus antibody at Screening and COVID-19 at Screening and Day -2.
* Willing to not consume citrus fruits (such as grapefruit, Seville oranges) and/or citrus fruit products throughout the study until Day 6.
* Willing to refrain from taking any prescription and non-prescription drugs, including herbal and nutritional supplements within 2 weeks prior to Day 1 and throughout the study until Day 6.
* CYP2D6 genotype that demonstrates gene variants of fast or intermediate metabolism (i.e. not ultra-rapid or poor).

Important Exclusion Criteria for both Stages 1 and 2:

* Current diagnosis of opioid or other substance dependence (except caffeine) according to DSM-IV or DSM-5 definitions (Stage 1 only).
* Any history of seizure or convulsion, including febrile convulsion in childhood or as an adult.
* History of chronic or frequent migraines.
* Current or recent (≤1 year) history of significant alcohol abuse (>3 units per day on a regular basis)
* For Stage 1, drug dependency disorder.
* For Stage 2, polydrug abuse or dependency within the past 3 years other than opioids, caffeine, and/or nicotine.
* Personal history or presence of primary psychotic disorder (including substance-induced or due to a medical condition), bipolar affective disorder Type I or Type II, or schizophrenia (not including non-psychotic, clinically stable disorders such as depression or anxiety).
* First or second-degree family history of primary psychotic disorder, bipolar affective disorder Type I or Type II, or schizophrenia.
* Showing suicidal tendency as per the Columbia Suicide Severity Rating Scale (C-SSRS).
* Any prior use of ibogaine, noribogaine or other chemically related substances or any allergy or intolerance to excipients in the ibogaine capsules.
* History or presence of clinically significant cardiovascular disease including angina, myocardial infarction, coronary artery disease, heart failure, arrhythmias, endocarditis, syncope of unknown origin, or any other condition that, in the opinion of the investigator, may be associated with a higher risk of arrhythmias.
* History or presence at screening (12-lead ECG and 24-hour Holter monitoring) or Day -2 (12-lead ECG) of ECGs that (1) shows QTcF interval duration >420 ms (if QTcF >420 ms prior to dosing on Day 1, subjects need not be excluded provided QTcF was ≤ 420 at Screening and Day -2 and QTcF ≤ 440 on Day 1.), PR interval duration >210 ms, or QRS interval duration >120 ms, obtained as an average from 3 ECG recordings, taken at least 1 minute apart after at least 10 minutes of quiet rest in the supine position; or (2) ECG showing ventricular bigeminy, trigeminy or couplets; or (3) shows, in the opinion of the investigator, any other clinically significant abnormality.
* History or family history of prolonged QT interval cardiac channelopathy or sudden cardiac death.
* Orthostatic hypotension or uncontrolled hypertension as characterized by sustained systolic elevation to ≥160 mmHg and/or diastolic elevation to ≥100 mmHg at screening or Day -2.
* Subjects with an average resting heart rate of <50 bpm on the ECG at screening.
* Use of any prescription drugs in the 28 days prior to the first study drug administration, that are known to inhibit or induce CYP2D6 or to cause QT prolongation or, in the opinion of the investigator, would put into question the status of the participant as healthy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
Stage 2 - Short Opiate Withdrawal Scale of Gossop (SOWS-Gossop) average score from Day 2 to Day 6 | Day 2 to Day 6
  The SOWS-Gossop is a 10-item questionnaire to evaluate opioid withdrawal symptom severity. Each item is scored on a 4-point scale. Higher scores indicate greater severity (total score range 0-40).

SECONDARY OUTCOMES:
Stage 2 - Subject completion status at Day 6 (key secondary endpoint) | Day 6
  Proportion of subjects who received study medication and completed the SOWS-Gossop assessment on Day 6
Stage 2 - Objective Opiate Withdrawal Scale of Handelsman (OOWS Handelsman) average score from Day 2 to Day 6 | Day 2 to Day 6
  The OOWS-Handelsman is an interview and observation tool for assessing opioid withdrawal signs and symptoms. It contains 13 physically observable signs, rated present or absent, based on a timed period of observation of the subject by a rater. Higher scores indicate greater severity (total score range 0-13).
Stage 2 - Subject completion status at Day 30 | Day 30
  Proportion of subjects who received study medication and completed the SOWS-Gossop assessment on Day 30
Stage 2 - Time to drop-out through Day 30 | Day 1 to Day 30
  Time to drop-out
Stage 2 - Daily subject-rated Visual Analog Scale for Efficacy (VAS-E) score from Day 2 to Day 6 and at Day 30 | Day 2 to Day 6 and at Day 30
  The VAS-E is a scale to quantify the state of craving a subject experienced in the previous 24 hours. The scale size is 100 mm, anchored on the left by "no craving at all" and anchored on the right by "strongest craving ever."
Stage 2 - Clinician-rated daily Clinical Global Impression - Improvement (CGI-I) score from Day 2 to Day 6 | Day 2 to Day 6
  The CGI-I is a 7-point scale that requires the clinician to assess how much the subject's condition has improved or worsened from baseline. The ratings are: 1 - very much improved; 2 - much improved; 3 - minimally improved; 4 - no change; 5 - minimally worse; 6 - much worse; 7 - very much worse.
Stage 2 - Hamilton Depression Rating Scale (HAM-D) score at Day 6 and Day 30 | Day 6 and Day 30
  The HAM-D is used to determine a subject's level of depression. The study uses the original 17-item scale. Higer scores indicate greater severity (total score range 0-52).
Stage 2 - Proportion of subjects requiring clonidine for relief of withdrawal symptoms up to Day 6 | Day 1 to Day 6
  Proportion of subjects requiring clonidine for relief of withdrawal symptoms

OTHER OUTCOMES:
Safety (Stage 1 and Stage 2) - Frequency of treatment-emergent adverse events | Day 1 to Day 30
  Number of subjects with treatment-emergent adverse events
Safety (Stage 1 and Stage 2) - number of subjects with abnormal electrocardiograms (ECG) | Day 1 to Day 30
  12-Lead ECG including heart rate (HR), QT interval corrected for HR according to Fridericia (QTcF), Individually corrected QTc interval (QTcI), HR-corrected J to T-peak interval (JTpc), PR interval, and QRS interval
Safety (Stage 1 and Stage 2) - number of subjects with new magnetic resonance imaging (MRI) findings (in the presence of ataxia greater than 24 hours post-dose) | Day 2
  MRI of the brain
Safety (Stage 1 and Stage 2) - number of subjects with abnormal neurological function | Day 2 to Day 6
  Neurological function
Safety (Stage 1 and Stage 2) - number of subjects with abnormal Scale for the Assessment and Rating of Ataxia (SARA) scores | Day 2
  The SARA is a tool for assessing ataxia. It includes 8 items related to gait, stance, sitting, speech, finger-chase test, nose-finger test, fast alternating movements and heel-shin test. Total scores range from 0 (no ataxia) to 40 (most severe ataxia).
Safety (Stage 2) - number of subjects with newly emerging suicidal ideation or behavior | Day 6 and Day 30
  Suicidality is assessed by means of the Columbia Suicide Severity Rating Scale (C-SSRS). It contains 6 "yes" or "no" questions (Q1: wish to be dead; Q2: non-specific suicidal thoughts; Q3-5: more specific suicidal thoughts and intent to act; Q6: suicidal behavior). An answer of "yes" to any of the six questions may indicate a need for referral to a trained mental health professional and an answer of "yes" to questions 4, 5 or 6 indicate high-risk.
Pharmacokinetics (Stage 1 and Stage 2) - maximum whole blood and plasma concentrations [Cmax] of ibogaine and noribogaine | 0.5 hours pre-dose up to 120 hours post-dose (Day 6)
  Whole blood and plasma concentrations
Pharmacokinetics (Stage 1 and Stage 2) - time to reach Cmax [Tmax] for ibogaine and noribogaine | 0.5 hours pre-dose up to 120 hours post-dose (Day 6)
  Tmax
Pharmacokinetics (Stage 1 and Stage 2) - area under the concentration-time curve up to the last measurable time point (AUC0-T) for ibogaine and noribogaine | 0.5 hours pre-dose up to 120 hours post-dose (Day 6)
  AUC0-T
Pharmacokinetics (Stage 1 and Stage 2) - apparent elimination half-life (T-half) of ibogaine and noribogaine | 0.5 hours pre-dose up to 120 hours post-dose (Day 6)
  T-half
Pharmacokinetics (Stage 1) - renal clearance (CLr) of ibogaine | 0.5 hours pre-dose up to 120 hours post-dose (Day 6)
  CLr

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - MAC Clinical Research Manchester (Early Phase Unit), Neuroscience Centre of Excellence, Manchester, Greater Mancherster
  - Hammersmith Medicines Research (HMR) Limited, London

IPD SHARING:
Plan to Share IPD: No